CLINICAL TRIAL: NCT00683007
Title: Use of Transesophageal Echocardiography to Assess Left Ventricular Performance During Acute Normovolemic Hemodilution and Randomized Replacement With Intravenous Crystalloid or Hypertonic Saline
Brief Title: Esophageal Echo Assessment of LV Function During Acute Normovolemic Hemodilution Using Crystalloid or Hypertonic Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 232664; 200815960 (Other: UC Davis Instructional Review Goard)
Record Dates: First submitted 2008-05-08; First posted 2008-05-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Hypovolemia
Keywords: TE echo; hemodilution; hypertonic; saline; Arterial Pressure Cardiac Output
MeSH Terms: interventions — Crystalloid Solutions; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Crystalloid
  Interventions: Other: Volume resuscitation (Crystalloid)
- 2 (Active Comparator): Hypertonic Saline
  Interventions: Other: Volume resuscitation (Hypertonic Saline Solution)

INTERVENTIONS:
Other: Volume resuscitation (Crystalloid) — Crystalloid vs. Hypertonic Saline Solution
  Arms: 1
Other: Volume resuscitation (Hypertonic Saline Solution) — Crystalloid vs. Hypertonic Saline Solution
  Arms: 2

SUMMARY:
The purpose of this study is to examine how the heart functions when a calculated amount of blood is removed and how two fluids, Lactated Ringer's (considered the standard replacement fluid) and Hypertonic Saline, re-expand the vascular system.

DETAILED DESCRIPTION:
This investigator-initiated, single-center, prospective, randomized, clinical experimental design will enroll 30 patients scheduled for elective radical prostatectomy, cystectomy, or cystoprostatectomy, and anterior/posterior spinal fusions, which includes routine acute normovolemic hemodilution (ANH) as a technique to decrease the need for banked blood transfusions. The purpose of this study is to compare two methods of volume replacement during the ANH procedure. Patients will be randomized to receive either standard crystalloid replacement with Lactated Ringers (LR) or 5% hypertonic saline. Selected measurements will be obtained by transesophageal echocardiography (TEE) for assessing changes in left ventricular volume and function associated with blood loss and replacement. This study will use the Accuson Cypress Cardiovascular System and the V5M transesophageal echocardiography probe (Siemens Medical Solutions, Malvern, PA). The TEE measurements will be recorded on magnetic optical discs and assessed off-line by the researcher after the data collection is completed using the proprietary software included in the ultrasound system. In addition, stroke volume variation measurement (SVV), Cardiac Output (CO), Cardiac Index (CI), and Stroke Volume Index (SVI) will be measured using the Vigileo (TM) arterial pressure monitor with the FloTrac (TM) sensor (Edwards Lifesciences, Irvine, CA).

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients requiring acute normovolemic hemodilution

Exclusion Criteria:

* Contraindication for hemodilution
* Contraindication for TE echo

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
TE echo LV 3-D volume changes. | 1 hour

SECONDARY OUTCOMES:
APCO system changes. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Neal W. Fleming, M.D., Ph.D., Study Director — Director, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine; David D. Rose, PhD, Principal Investigator — Chief, Certified Registered Nurse Anesthetist, UC Davis, Department of Anesthesiology and Pain Medicine
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Cheung AT, Savino JS, Weiss SJ, Aukburg SJ, Berlin JA. Echocardiographic and hemodynamic indexes of left ventricular preload in patients with normal and abnormal ventricular function. Anesthesiology. 1994 Aug;81(2):376-87. doi: 10.1097/00000542-199408000-00016. PMID 8053588
- [Background] Kungys G, Rose DD, Fleming NW. Stroke volume variation during acute normovolemic hemodilution. Anesth Analg. 2009 Dec;109(6):1823-30. doi: 10.1213/ANE.0b013e3181ba41af. PMID 19923509